CLINICAL TRIAL: NCT01810913
Title: Randomized Phase II/III Trial of Adjuvant Radiation Therapy With Cisplatin, Docetaxel-Cetuximab, or Cisplatin-Atezolizumab in Pathologic High-Risk Squamous Cell Cancer of the Head and Neck
Brief Title: Testing Docetaxel-Cetuximab or the Addition of an Immunotherapy Drug, Atezolizumab, to the Usual Chemotherapy and Radiation Therapy in High-Risk Head and Neck Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00500; NCI-2013-00500 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG-1216 (Other: NRG Oncology); RTOG-1216 (Other: CTEP); U10CA021661 (NIH); U10CA180868 (NIH); NCT04411121 (obsolete NCT alias)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Oropharyngeal p16INK4a-Negative Squamous Cell Carcinoma; Stage III Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage III Laryngeal Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7; Stage IV Hypopharyngeal Squamous Cell Carcinoma AJCC v7; Stage IV Laryngeal Squamous Cell Carcinoma AJCC v7; Stage IV Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IV Oropharyngeal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — atezolizumab; Biopsy; Specimen Handling; Cetuximab; (225)Ac-DOTA-c(RGDyK); Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (IMRT, cisplatin) (Experimental): Patients undergo IMRT QD five days a week for 6 weeks and receive concurrent cisplatin IV over 1-2 hours once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo collection of blood samples during screening and throughout the study and may undergo CT scans and/or MRI and biopsy as clinically indicated on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Other: Survey Administration
- Arm 2 (IMRT, docetaxel) (Experimental): Patients undergo IMRT as in Arm I and receive concurrent docetaxel IV over 60 minutes once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo CT scans and/or MRI, and collection of blood during follow-up. (CLOSED AS OF 20-MAR-2020)
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Docetaxel; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Other: Survey Administration
- Arm 3 (IMRT, docetaxel, cetuximab) (Experimental): Patients receive cetuximab IV over 120 minutes on week 1 and over 60 minutes once weekly on weeks 2-7. Patients undergo IMRT as in Arm I and receive concurrent docetaxel once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo collection of blood samples during screening and throughout the study and may undergo CT scans and/or MRI and biopsy as clinically indicated on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Biological: Cetuximab; Procedure: Computed Tomography; Drug: Docetaxel; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Other: Survey Administration
- Arm 4 (IMRT, cisplatin, atezolizumab) (Experimental): Patients undergo IMRT QD five days a week for 6 weeks and receive concurrent cisplatin IV over 1-2 hours once weekly for 6 weeks. Starting 1 week before IMRT, patients also receive atezolizumab IV over 30-60 minutes every 3 weeks for up to 8 doses (weeks -1, 3, 6, 9, 12, 15, 18, and 21) in the absence of disease progression and unacceptable toxicity. Patients undergo collection of blood samples during screening and throughout the study and may undergo CT scans and/or MRI and biopsy as clinically indicated on study.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Other: Survey Administration

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm 4 (IMRT, cisplatin, atezolizumab)
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Arm 1 (IMRT, cisplatin); Arm 3 (IMRT, docetaxel, cetuximab); Arm 4 (IMRT, cisplatin, atezolizumab)
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cetuximab — Given IV
  Other Names: C 225; C-225; C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm 3 (IMRT, docetaxel, cetuximab)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm 1 (IMRT, cisplatin); Arm 4 (IMRT, cisplatin, atezolizumab)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm 2 (IMRT, docetaxel); Arm 3 (IMRT, docetaxel, cetuximab)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II/III trial studies how well radiation therapy works when given together with cisplatin, docetaxel, cetuximab, and/or atezolizumab after surgery in treating patients with high-risk stage III-IV head and neck cancer the begins in the thin, flat cells (squamous cell). Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as cisplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cetuximab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The purpose of this study is to compare the usual treatment (radiation therapy with cisplatin chemotherapy) to using radiation therapy with docetaxel and cetuximab chemotherapy, and using the usual treatment plus an immunotherapy drug, atezolizumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To select the better docetaxel-based experimental arm to improve disease-free survival (DFS) over the control arm of radiation and cisplatin. (Phase II) (COMPLETE AS OF 20-MAR-2020) II. To determine if the combination of docetaxel-cetuximab and intensity-modulated radiation therapy (IMRT) is superior in terms of overall survival (OS) compared to standard cisplatin and IMRT in the adjuvant treatment of pathologic high risk, human papillomavirus (HPV)-negative head and neck squamous cell carcinoma (HNSCC). (Phase III) III. To determine if the combination of atezolizumab, cisplatin, and IMRT is superior in terms of OS compared to standard cisplatin and IMRT in the adjuvant treatment of pathologic high risk, HPV-negative HNSCC. (Phase III)

SECONDARY OBJECTIVES:

I. To compare disease-free survival (DFS) between each experimental arm and the control arm. (Phase III) II. To determine whether each experimental arm improves local-regional disease control and the rate of distant metastasis. (Phase III) III. To compare acute toxicity profiles between each experimental arm and the control arm. (Phase III) IV. To compare late toxicity profiles at 1, 3, and 5 years after treatment. (Phase III) V. To assess long term DFS and OS between each experimental arm and the control arm. (Phase III) VI. To compare symptom burden, as measured by the MD Anderson Symptom Inventory - Head and Neck (MDASI-HN) (primary patient reported outcome [PRO]), and quality of life, as measured by the Functional Assessment of Cancer Therapy - Head and Neck (FACT-H&N) (secondary PRO), between each experimental arm and the control arm. (Phase III)

EXPLORATORY OBJECTIVE:

I. To collect blood and tissue specimens for future translational research. (Phase III)

OUTLINE: Patients are randomized to 1 of 3 arms - Phase II (Arms 1, 2 or 3) and for Phase III (Arms 1, 3 or 4).

ARM 1: Patients undergo intensity modulated radiation therapy (IMRT) once daily (QD) five days a week for 6 weeks and receive concurrent cisplatin intravenously (IV) over 1-2 hours once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients undergo IMRT as in Arm I and receive concurrent docetaxel IV over 60 minutes once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity. (CLOSED AS OF 20-MAR-2020)

ARM 3: Patients receive cetuximab IV over 120 minutes on week 1 and over 60 minutes once weekly on weeks 2-7. Patients undergo IMRT as in Arm I and concurrently receive docetaxel once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM 4: Patients undergo IMRT QD five days a week for 6 weeks and receive concurrent cisplatin IV over 1-2 hours once weekly for 6 weeks. Starting 1 week before IMRT, patients also receive atezolizumab IV over 30-60 minutes every 3 weeks for up to 8 doses (weeks -1, 3, 6, 9, 12, 15, 18, and 21) in the absence of disease progression and unacceptable toxicity.

All patients undergo collection of blood samples during screening and throughout the study and may undergo computed tomography (CT) scans and/or magnetic resonance imaging (MRI) and biopsy as clinically indicated on study.

After completion of study treatment, patients are followed up at 1 and 3 months, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PHASE II INCLUSION CRITERIA (COMPLETE AS OF 20-MAR-2020)
* Pathologically (histologically or cytologically) proven diagnosis of head and neck squamous cell carcinoma (HNSCC) involving the oral cavity (excluding lips), oropharynx (p16 negative), larynx, or hypopharynx
* Patients must have undergone gross total surgical resection of high-risk oral cavity, oropharynx (p16 negative), larynx, or hypopharynx within 63 days prior to registration; Note: patients may have biopsy under general anesthesia in an operating room followed by definitive ablative cancer surgery representing gross total resection; the gross total resection has to be done within 63 days prior to registration; if, however, patients have ablative resection but shortly recur or are determined to have persisting disease requiring re-resection to achieve gross total resection, then the patient is not eligible
* Patients must have at least 1 of the following high-risk pathologic features: extracapsular nodal extension or invasive cancer at the primary tumor resection margin (tumor on ink)
* Pathologic stage III or IV HNSCC, including no distant metastases, based upon the following minimum diagnostic workup:

  * General history and physical examination by a radiation oncologist and/or medical oncologist within 84 days prior to registration;
  * Examination by an ear nose throat (ENT) or head & neck surgeon prior to surgery; a laryngopharyngoscopy (mirror and/or fiber optic and/or direct procedure), if appropriate, is recommended but not required; intra-operative examination is acceptable documentation
  * Pre-operative (op) Imaging of the head and neck: A neck computed tomography (CT) (with contrast) or CT/positron emission tomography (PET) (with contrast) and/or an magnetic resonance imaging (MRI) of the neck (T1 with gadolinium and T2) within 84 days prior to surgery; Note: this imaging data (diagnostic pre-operative scan showing gross disease) is to be submitted in Digital Imaging and Communications in Medicine (DICOM) format via TRIAD; the report is to be uploaded into Rave
  * Chest CT scan (with or without contrast) or CT/PET that includes the chest (with or without contrast) either within 84 days prior to surgery or within 120 days prior to registration; Note: if the CT/PET with or without contrast is done within 84 days prior to surgery, it fulfills the chest imaging requirement
* Zubrod performance status of 0-1 within 14 days prior to registration
* Age >= 18
* Absolute granulocyte count (AGC) >= 1,500 cells/mm^3 (obtained within 14 days prior to registration on study)
* Platelets >= 100,000 cells/mm^3 (obtained within 14 days prior to registration on study)
* Hemoglobin >= 8.0 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Total bilirubin < 2 x institutional upper limit of normal (ULN) within 14 days prior to registration
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x institutional ULN within 14 days prior to registration
* Serum creatinine institutional ULN within 14 days prior to registration or; creatinine clearance (CC) >= 50 ml/min within 14 days prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula
* Negative urine or serum pregnancy test within 14 days prior to registration for women of childbearing potential
* The following assessments are required within 14 days prior to registration: sodium (Na), potassium (K), chloride (Cl), glucose, calcium (Ca), magnesium (Mg), and albumin; Note: patients with an initial magnesium < 0.5 mmol/L (1.2 mg/dl) may receive corrective magnesium supplementation but should continue to receive either prophylactic weekly infusion of magnesium and/or oral magnesium supplementation (e.g., magnesium oxide) at the investigator's discretion
* Patients with feeding tubes are eligible for the study
* Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control
* Patient must provide study specific informed consent prior to study entry, including consent for mandatory tissue submission for epidermal growth factor receptor (EGFR) analysis and for oropharyngeal cancer patients, human papilloma virus (HPV) analysis
* PHASE III: Pathologically (histologically or cytologically) proven diagnosis of head and neck squamous cell carcinoma (HNSCC) involving the oral cavity (excluding lips), oropharynx (p16 negative), larynx, or hypopharynx
* PHASE III: Patients with oropharyngeal cancer must have p16-negative based on central review prior to Step 2 registration. All patients with oropharyngeal primary must consent for mandatory tissue submission for central p16 confirmation
* PHASE III: Patients must have undergone gross total surgical resection of high-risk oral cavity, oropharynx (p16 negative), larynx, or hypopharynx within 63 days prior to registration

  * Note: Patients may have biopsy under general anesthesia in an operating room followed by definitive ablative cancer surgery representing gross total resection. The gross total resection has to be done within 63 days prior to registration. If, however, patients have ablative resection but shortly recur or are determined to have persisting disease requiring re-resection to achieve gross total resection, then the patient is not eligible
* PHASE III: Patients must have at least 1 of the following high-risk pathologic features: extracapsular nodal extension or invasive cancer at the primary tumor resection margin (tumor on ink or tumor in a final separately submitted margin)
* PHASE III: Pathologic stage III or IV HNSCC (American Joint Committee on Cancer [AJCC] 7th edition), including no distant metastases, based upon the following minimum diagnostic workup:

  * General history and physical examination by a radiation oncologist or medical oncologist within 84 days prior to registration;
  * Examination by an ENT or head & neck surgeon prior to surgery; a laryngopharyngoscopy (mirror or fiberoptic or direct procedure), if appropriate, is recommended but not required. Intra-operative examination is acceptable documentation.
  * Pre-op Imaging of the head and neck: A neck CT (with contrast and of diagnostic quality) or PET/CT (with contrast and of diagnostic quality) and/or an MRI of the neck of diagnostic quality (T1 with gadolinium and T2) within 84 days prior to surgery; Note: this imaging data (diagnostic pre-operative scan showing gross disease) is to be submitted in DICOM format via TRIAD. The report is to be uploaded into Rave.
  * Chest CT scan (with or without contrast) or PET/CT that includes the chest (with or without contrast) either within 84 days prior to surgery or within 120 days prior to registration; Note: If the PET/CT with or without contrast is done within 84 days prior to surgery, it fulfills the chest imaging requirement
* PHASE III: Zubrod performance status of 0-1 within 14 days prior to registration
* PHASE III: Age >= 18
* PHASE III: Leukocytes >= 2,500 cells/mm^3 (obtained within 14 days prior to registration on study)
* PHASE III: Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (obtained within 14 days prior to registration on study)
* PHASE III: Platelets >= 100,000 cells/mm^3 (obtained within 14 days prior to registration on study)
* PHASE III: Hemoglobin >= 8.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb >= 8.0 g/dL is acceptable) (obtained within 14 days prior to registration on study)
* PHASE III: Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x institutional ULN may be enrolled) (within 14 days prior to registration)
* PHASE III: AST or ALT =< 3 x institutional ULN (within 14 days prior to registration)
* PHASE III: Alkaline phosphatase =< 2.5 x institutional ULN (within 14 days prior to registration)
* PHASE III: Creatinine clearance (CrCl) >= 50 mL/min within 14 days prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula
* PHASE III: Patients with feeding tubes are eligible for the study
* PHASE III: Negative urine or serum pregnancy test within 14 days prior to registration for women of childbearing potential
* PHASE III: All patients must provide study specific informed consent prior to study entry
* PHASE III: Patients positive for human immunodeficiency virus (HIV) are allowed on study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART);
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections;
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based tests

Exclusion Criteria:

* PHASE II EXCLUSION CRITERIA (COMPLETE AS OF 20-MAR-2020)
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years); noninvasive cancers (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible) are permitted even if diagnosed and treated < 3 years ago
* Patients with simultaneous primaries or bilateral tumors are excluded, with the exception of patients with bilateral tonsil cancers or patients with T1-2, N0, M0 resected differentiated thyroid carcinoma, who are eligible
* Prior systemic chemotherapy or anti-epidermal growth factor (EGF) therapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within 6 months prior to registration
  * Transmural myocardial infarction within 6 months prior to registration
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration

    * Idiopathic pulmonary fibrosis or other severe interstitial lung disease that requires oxygen therapy or is thought to require oxygen therapy within 1 year prior to registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol

    * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease and Control and Prevention (CDC) definition; note: human immunodeficiency virus (HIV) testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive; protocol-specific requirements may also exclude immuno-compromised patients.
* Grade 3-4 electrolyte abnormalities (Common Terminology Criteria for Adverse Events [CTCAE], version [v.] 4):
* Serum calcium (ionized or adjusted for albumin) < 7 mg/dl (1.75 mmol/L) or > 12.5 mg/dl (> 3.1 mmol/L) despite intervention to normalize levels
* Glucose < 40 mg/dl (< 2.2 mmol/L) or > 250 mg/dl (> 14 mmol/L)
* Magnesium < 0.9 mg/dl (< 0.4 mmol/L) or > 3 mg/dl (> 1.23 mmol/L) despite intervention to normalize levels
* Potassium < 3.0 mmol/L or > 6 mmol/L despite intervention to normalize levels
* Sodium < 130 mmol/L or > 155 mmol/L despite intervention to normalize levels
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Prior allergic reaction to cetuximab
* PHASE III: Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years) with the following exceptions: T1-2, N0, M0 resected differentiated thyroid carcinoma; Note that noninvasive cancers (For example, carcinoma in situ of the breast, oral cavity, or cervix) are permitted even if diagnosed and treated < 3 years ago
* PHASE III: Patients with simultaneous primaries or bilateral tumors are excluded, with the exception of patients with bilateral tonsil cancers or patients with T1-2, N0, M0 resected differentiated thyroid carcinoma, who are eligible
* PHASE III: Prior systemic therapy, including cytotoxic chemotherapy, biologic/targeted therapy (such as anti-EGF therapy), or immune therapy for the study cancer; note that prior chemotherapy for a different cancer is allowable, however, a prior anti-PD-1, anti-PD-L1, or anti-PD-L2 agent is not permitted
* PHASE III: Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* PHASE III: Severe, active co-morbidity, defined as follows:

  * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification; to be eligible for this trial, patients should be class 2B or better within 6 months prior to registration
  * Transmural myocardial infarction within 6 months prior to registration;
  * Severe infections within 4 weeks prior to registration including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia;
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; Note: Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible.
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
  * History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in a prior radiation field (fibrosis) is permitted, provided that field does not overlap with the planned radiation field for the study cancer;
  * Patients with active tuberculosis (TB) are excluded;
  * Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease;

    * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
  * History of allogeneic bone marrow transplantation or solid organ transplantation.
  * A diagnosis of immunodeficiency:

    * Acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note: HIV testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
  * Is receiving treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to registration.

    * Note: Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
    * Note: The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
  * History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

    * Patients with a history of autoimmune hypothyroidism who are asymptomatic and/or are on a stable dose of thyroid replacement hormone are eligible.
    * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* PHASE III: Grade 3-4 electrolyte abnormalities (CTCAE, v. 4) within 14 days prior to registration:

  * Serum calcium (ionized or adjusted for albumin) < 7 mg/dL (1.75 mmol/L) or > 12.5 mg/dL (> 3.1 mmol/L) despite intervention to normalize levels;
  * Glucose < 40 mg/dL (< 2.2 mmol/L) or > 250 mg/dL (> 14 mmol/L);
  * Magnesium < 0.9 mg/dL (< 0.4 mmol/L) or > 3 mg/dL (> 1.23 mmol/L) despite intervention to normalize levels;
  * Potassium < 3.0 mmol/L or > 6 mmol/L despite intervention to normalize levels;
  * Sodium < 130 mmol/L or > 155 mmol/L despite intervention to normalize levels.
* PHASE III: Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception for up to 5 months from last study treatment; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic. Women who are breastfeeding and unwilling to discontinue are also excluded
* PHASE III: History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* PHASE III: Patients taking bisphosphonate therapy for symptomatic hypercalcemia. Use of bisphosphonate therapy for other non-oncologic reasons (e.g., osteoporosis) is allowed
* PHASE III: Patients requiring treatment with a RANKL inhibitor (e.g. denosumab) for non-oncologic reasons who cannot discontinue it before registration
* PHASE III: Patients with known distant metastatic disease are excluded
* PHASE III: Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* PHASE III: Major surgical procedure within 28 days prior to registration or anticipation of need for a major surgical procedure during the course of the study
* PHASE III: Administration of a live, attenuated vaccine within 4 weeks prior to registration or anticipation that such a live, attenuated vaccine will be required during the study and for patients receiving atezolizumab, up to 5 months after the last dose of atezolizumab.

  * Influenza vaccination should be given during influenza season only (approximately October to

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Estimated)
Dates: Start 2013-03-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (Phase II) | From date of randomization until date of local-regional recurrence, distant metastasis or death due to any cause, assessed up to 7 years
  Estimated using the Kaplan-Meier method for each arm. Their distributions will be compared between treatment arms with a one-sided log rank test.
Overall survival (Phase III) | From date of randomization to death due to any cause, assessed up to 7 years
  Estimated using the Kaplan-Meier method for each arm. Their distributions will be compared between treatment arms with a one-sided log rank test. Multivariate analysis will be performed using the Cox proportional hazards model.

SECONDARY OUTCOMES:
Local-regional failure | From date of randomization until date of local-regional recurrence, assessed up to 7 years
  The cumulative incidence method will be used to estimate rates, and the failure rates for the experimental arms will be compared against the control using a failure-specific log rank test.
Distant metastasis | From date of randomization to date of distant metastasis, assessed up to 7 years
  The cumulative incidence method will be used to estimate rates, and the failure rates for the experimental arms will be compared against the control using a failure-specific log rank test.
Toxicity | From start of treatment to death or last follow-up
  Adverse events will be graded using Common Terminology Criteria for Adverse Events version 4.0. Rates of grade 3+ adverse events overall will be compared between arms by Chi-square test, or Fisher's exact test.
Patient-reported outcome, symptom burden | Time from randomization to a first recovery within at least one MID unit of total symptom severity compared to the baseline (reference) score
  Time to recovery of baseline total symptom severity from the MD Anderson Symptom Inventory - Head and Neck. The cumulative incidence method will be used to estimate the event rates, and the event rates between arms will be compared using a cause-specific log rank test. The Fine-Gray subdistribution hazards model may be applied to further explore outcomes by treatment arm and other covariates.
Quality of life | Baseline and 1 year post radiation therapy
  Quality of life change from baseline at 1-year post RT, as measured by the Functional Assessment of Cancer Therapy - Head and Neck (FACT) Trial Outcome Index (TOI). FACT TOI is a validated efficient summary index of physical/functional outcomes, and disease site-specific items, which is highly reliable and sensitive to change in performance status rating. A constrained longitudinal data analysis model will be fitted with all the time points (discrete), the treatment factor and its interaction. The secondary non-inferiority patient-reported outcome hypothesis will be tested using a confidence interval approach.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Harari, Principal Investigator — NRG Oncology
Locations (336):
- United States (332):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Saint Helena Hospital, St. Helena, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center at SouthShore, Ruskin, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Ascension Saint Vincent Anderson, Anderson, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - South Shore University Hospital, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - East Carolina University, Greenville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Saint Francis Hospital, Federal Way, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Spokane Valley Cancer Center-Mission, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong